CLINICAL TRIAL: NCT00250432
Title: A Multicenter, Randomized, Double-Blind, Comparative Study to Evaluate the Safety, Tolerability, and Efficacy of 2 Dosing Regimens of Caspofungin in the Treatment of Invasive Candidiasis in Adults
Brief Title: A Multicenter, Randomized, Double-Blind, Comparative Study to Evaluate the Safety, Tolerability, and Efficacy of 2 Dosing Regimens of an Antifungal Drug in the Treatment of Fungal Infections in Adults (0991-801)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0991-801; 2005_085
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Results first posted 2009-03-24 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Invasive Candidiasis
MeSH Terms: conditions — Candidiasis, Invasive | interventions — Caspofungin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): 50 mg intravenous (IV) infusion (diluted with 9% saline) administered daily (following a 70-mg IV loading dose on Day 1), over the course of ~2 hrs. all patients should be treated with antifungal therapy for at least 14 days following both the improvement in clinical and radiographic signs of disease and the eradication of Candida from culture samples obtained from the invasive site of infection.
  Interventions: Drug: caspofungin acetate
- 2 (Experimental): 150 mg intravenous (IV) infusion (diluted with 9% saline) administered daily, over the course of ~2 hrs. all patients should be treated with antifungal therapy for at least 14 days following both the improvement in clinical and radiographic signs of disease and the eradication of Candida from culture samples obtained from the invasive site of infection.
  Interventions: Drug: caspofungin acetate

INTERVENTIONS:
Drug: caspofungin acetate — Caspofungin acetate 50 mg IV infusion (diluted with 9% saline) (following a 70-mg IV loading dose on Day 1); Caspofungin acetate 150 mg IV infusion (diluted with 9% saline) administered daily, over the course of ~2 hrs. Duration of Treatment - 14-90 days.

SUMMARY:
Comparison of the safety and effectiveness of standard drug dosing versus a daily dose 3 times higher than the standard dose in patients with invasive candidiasis (bloodstream and/or systemic yeast infections)

ELIGIBILITY:
Inclusion Criteria:

* Clinical and Laboratory evidence of blood stream &/or systemic candida infections

Exclusion Criteria:

* Possible candida contamination
* Candida colonization (non invasive infection), urine, cardiac, bone or brain and prosthetic device infections
* Acute or moderately severe liver disease
* Abnormal liver function tests
* Abnormal blood clotting for patients on blood thinners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Betts RF, Nucci M, Talwar D, Gareca M, Queiroz-Telles F, Bedimo RJ, Herbrecht R, Ruiz-Palacios G, Young JA, Baddley JW, Strohmaier KM, Tucker KA, Taylor AF, Kartsonis NA; Caspofungin High-Dose Study Group. A Multicenter, double-blind trial of a high-dose caspofungin treatment regimen versus a standard caspofungin treatment regimen for adult patients with invasive candidiasis. Clin Infect Dis. 2009 Jun 15;48(12):1676-84. doi: 10.1086/598933. PMID 19419331

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase III study. The first patient was enrolled (FPE) on 13-Jan-2006. The last patient's last visit (LPLV) was on 13-Mar-2008. A total of 38 inpatient centers were involved in the recruitment worldwide (14 in the United States, 13 in the European Union, 7 in Central or South America, and 4 in Asia)
Groups:
- Caspofungin 70/50 mg: Caspofungin 50 mg IV daily (following a 70-mg IV loading dose on Day 1)
- Caspofungin 150 mg: Caspofungin 150 mg IV daily
Period: Overall Study
Arm/Group | Caspofungin 70/50 mg | Caspofungin 150 mg
Started | 104 | 100
Completed | 59 | 53
Not Completed | 45 | 47
Not completed — Adverse Event | 25 | 29
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 6 | 5
Not completed — Patient Moved | 0 | 1
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Pt died out of posttherapy report period | 6 | 5
Not completed — Pt was considered untreatable | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caspofungin 70/50 mg | Caspofungin 150 mg | Total
Number analyzed (Participants) | 104 | 100 | 204
Age, Continuous [Mean (Full Range); unit: years] | 56.0 [16 to 90] | 57.8 [20 to 87] | 56.9 [16 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 40 | 90
  Male | 54 | 60 | 114
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 70 | 65 | 135
  Black | 11 | 12 | 23
  Asian | 17 | 16 | 33
  Hispanic | 4 | 5 | 9
  Other | 2 | 2 | 4
Site Of Invasive Candida Infection [Number; unit: Participants] — This table lists the site of invasive candidiasis. Patients are included in only 1 category. Patients with more than 1 site of infection are counted under "Acute disseminated candidiasis or multiple sites".
  Participants
    Abscess(involving an intra-abdominal site) | 0 | 2 | 2
    Abscess (involving a non-abdominal site) | 0 | 1 | 1
    Acute disseminated candidiasis or multiple sites | 6 | 7 | 13
    Blood (candidemia) | 91 | 81 | 172
    Chronic disseminated candidiasis (hepatosplenic) | 1 | 0 | 1
    Fungemia (non Candida) | 0 | 2 | 2
    Kidney (Pyelonephritis) | 0 | 1 | 1
    Lung (Pneumonia) | 1 | 1 | 2
    Peritoneal fluid (Peritonitis) | 4 | 5 | 9
    Pleural fluid (Empyema) | 1 | 0 | 1
APACHE II Score (at Study Entry) [Mean (Full Range); unit: Units on a Scale] — APACHE (Acute Physiology and Chronic Health Evaluation) is a system of classifying severity of illnesses in intensive care patients. The possible range of values is 0 (minimum severity) to 71 (maximum severity).
  Units on a Scale | 16.5 [3 to 38] | 17.0 [2 to 39] | 16.8 [2 to 39]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Develop Significant Drug-related Adverse Events.
Description: Number of patients with at least 1 significant drug-related adverse event (serious drug-related or drug-related adverse events leading to caspofungin discontinuation) while on caspofungin study therapy or during the immediate 14-day post-caspofungin therapy period.
Time Frame: 90 Days
Population: All patients as treated population
Measure: Number; unit: Participants
Arm/Group | Caspofungin 70/50 mg | Caspofungin 150 mg
Number analyzed (Participants) | 104 | 100
Participants | 2 | 3
Statistical Analysis 1: Comparison: Caspofungin 70/50 mg vs Caspofungin 150 mg; A significant drug-related adverse event was defined as either a drug-related serious adverse event or a drug-related adverse event leading to discontinuation of caspofungin therapy. Comparison between the 2 caspofungin groups was based on upper bound of the 95% confidence interval for the difference; Test type: Non-Inferiority or Equivalence — Safety with caspofungin 150 mg daily will be non-inferior to that of caspofungin 70/50 mg. Non-inferiority was defined as upper limit of the 2-sided, 95% confidence interval for the difference (150-mg group - 70/50-mg group) must be less than 0.15 (15 percentage points); Rate Difference = 1.1, 95% CI [-4.1 to 6.8], Standard Error of Mean 5.6 — The confidence interval computation was based on the method by Miettinen and Nurminen

2. Secondary Outcome: Number of Patients With a Favorable Overall Response.
Description: Number of patients with a favorable overall response, defined as a clinical response of "cure" or "apparent cure" along with a microbiological response of "eradication" or "presumptive eradication" at the End of Caspofungin Therapy.
Time Frame: 90 Days
Population: Full Analysis Set (FAS): Included those patients who received at least 1 full dose of caspofungin study therapy and had a documented diagnosis of invasive candidiasis from a sterile, invasive body site, as defined in the protocol.
Measure: Number; unit: Participants
Arm/Group | Caspofungin 70/50 mg | Caspofungin 150 mg
Number analyzed (Participants) | 102 | 95
Participants | 73 | 74
Statistical Analysis 1: Comparison: Caspofungin 70/50 mg vs Caspofungin 150 mg; There was no formal hypothesis testing for efficacy in this study. The main efficacy analysis was the number (percentage) of patients with a favorable overall response at the end of caspofungin study therapy, together with the within treatment 95% exact binomial confidence intervals, and the estimated treatment difference, and its 95% confidence interval; Test type: Superiority or Other; Rate Difference = 6.3, 95% CI [-5.9 to 18.4], Standard Error of Mean 12.1 — The 95% confidence interval on the difference will be based on the method of Miettinen and Nurminen

ADVERSE EVENTS:
Arm/Group | Caspofungin 70/50 mg | Caspofungin 150 mg
Serious Adverse Events (participants affected / at risk) | 46 | 44
Other Adverse Events (participants affected / at risk) | 69 | 70
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Caspofungin 70/50 mg | Caspofungin 150 mg
Leukopenia (Blood and lymphatic system disorders) | 0/104 | 1/100
Acute Myocardial Infarction (Cardiac disorders) | 1/104 | 0/100
Arrhythmia (Cardiac disorders) | 0/104 | 1/100
Atrioventricular Block (Cardiac disorders) | 0/104 | 1/100
Atrioventricular Block Complete (Cardiac disorders) | 1/104 | 0/100
Bradycardia (Cardiac disorders) | 0/104 | 1/100
Cardiac Arrest (Cardiac disorders) | 1/104 | 1/100
Cardiac Failure Congestive (Cardiac disorders) | 0/104 | 1/100
Cardio-Respiratory Arrest (Cardiac disorders) | 2/104 | 0/100
Electromechanical Disorder (Cardiac disorders) | 1/104 | 0/100
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1/104 | 1/100
Gastrointestinal Ulcer Perforation (Gastrointestinal disorders) | 0/104 | 1/100
Haematemesis (Gastrointestinal disorders) | 1/104 | 0/100
Intestinal Obstruction (Gastrointestinal disorders) | 0/104 | 1/100
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 0/104 | 1/100
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1/104 | 0/100
Peritoneal Haemorrhage (Gastrointestinal disorders) | 0/104 | 1/100
Vomiting (Gastrointestinal disorders) | 1/104 | 0/100
Brain Death (General disorders) | 1/104 | 0/100
Death (General disorders) | 2/104 | 0/100
General Physical Health Deterioration (General disorders) | 1/104 | 0/100
Multi-Organ Failure (General disorders) | 5/104 | 4/100
Non-Cardiac Chest Pain (General disorders) | 1/104 | 0/100
Pyrexia (General disorders) | 1/104 | 0/100
Systemic Inflammatory Response Syndrome (General disorders) | 0/104 | 1/100
Hepatitis Toxic (Hepatobiliary disorders) | 0/104 | 1/100
Hyperbilirubinaemia (Hepatobiliary disorders) | 0/104 | 1/100
Jaundice Cholestatic (Hepatobiliary disorders) | 1/104 | 0/100
Abdominal Sepsis (Infections and infestations) | 0/104 | 2/100
Bacteraemia (Infections and infestations) | 2/104 | 0/100
Cellulitis (Infections and infestations) | 2/104 | 0/100
Cholecystitis Infective (Infections and infestations) | 0/104 | 1/100
Clostridial Infection (Infections and infestations) | 1/104 | 0/100
Enterococcal Bacteraemia (Infections and infestations) | 0/104 | 2/100
Fungaemia (Infections and infestations) | 2/104 | 0/100
Fungal Sepsis (Infections and infestations) | 0/104 | 1/100
Klebsiella Bacteraemia (Infections and infestations) | 0/104 | 1/100
Lower Respiratory Tract Infection (Infections and infestations) | 0/104 | 1/100
Meningitis Aseptic (Infections and infestations) | 1/104 | 0/100
Pneumonia (Infections and infestations) | 3/104 | 4/100
Pneumonia Staphylococcal (Infections and infestations) | 1/104 | 0/100
Pseudomonal Bacteraemia (Infections and infestations) | 0/104 | 1/100
Sepsis (Infections and infestations) | 5/104 | 6/100
Septic Shock (Infections and infestations) | 12/104 | 13/100
Stenotrophomonas Infection (Infections and infestations) | 0/104 | 1/100
Systemic Candida (Infections and infestations) | 1/104 | 1/100
Urosepsis (Infections and infestations) | 0/104 | 1/100
Wound Infection (Infections and infestations) | 1/104 | 0/100
Accidental Overdose (Injury, poisoning and procedural complications) | 0/104 | 1/100
Tracheal Obstruction (Injury, poisoning and procedural complications) | 0/104 | 1/100
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0/104 | 1/100
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/104 | 1/100
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/104 | 0/100
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/104 | 1/100
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/104 | 0/100
Pituitary Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/104 | 0/100
Tumour Necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/104 | 0/100
Cerebral Haematoma (Nervous system disorders) | 1/104 | 0/100
Convulsion (Nervous system disorders) | 2/104 | 0/100
Myasthenia Gravis (Nervous system disorders) | 0/104 | 1/100
Partial Seizures (Nervous system disorders) | 0/104 | 1/100
Oliguria (Renal and urinary disorders) | 0/104 | 1/100
Renal Failure Acute (Renal and urinary disorders) | 2/104 | 2/100
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1/104 | 0/100
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2/104 | 3/100
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1/104 | 1/100
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1/104 | 0/100
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0/104 | 1/100
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0/104 | 1/100
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1/104 | 0/100
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1/104 | 1/100
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0/104 | 1/100
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 2/104 | 1/100
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0/104 | 1/100
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6/104 | 1/100
Haemodynamic Instability (Vascular disorders) | 0/104 | 1/100
Peripheral Vascular Disorder (Vascular disorders) | 0/104 | 1/100
Shock Haemorrhage (Vascular disorders) | 0/104 | 1/100
Venous Thrombosis Limb (Vascular disorders) | 1/104 | 0/100
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Caspofungin 70/50 mg | Caspofungin 150 mg
Anaemia (Blood and lymphatic system disorders) | 3/104 | 4/100
Atrial Fibrillation (Cardiac disorders) | 0/104 | 3/100
Bradycardia (Cardiac disorders) | 2/104 | 2/100
Tachycardia (Cardiac disorders) | 1/104 | 2/100
Ventricular Tachycardia (Cardiac disorders) | 3/104 | 2/100
Adrenal Insufficiency (Endocrine disorders) | 0/104 | 2/100
Abdominal Pain (Gastrointestinal disorders) | 3/104 | 0/100
Abdominal Pain Upper (Gastrointestinal disorders) | 2/104 | 3/100
Constipation (Gastrointestinal disorders) | 3/104 | 3/100
Diarrhea (Gastrointestinal disorders) | 6/104 | 7/100
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1/104 | 2/100
Haematemesis (Gastrointestinal disorders) | 0/104 | 2/100
Ileus (Gastrointestinal disorders) | 3/104 | 1/100
Nausea (Gastrointestinal disorders) | 5/104 | 7/100
Vomiting (Gastrointestinal disorders) | 10/104 | 6/100
Asthenia (General disorders) | 2/104 | 3/100
Chest Pain (General disorders) | 1/104 | 2/100
Generalised Oedema (General disorders) | 3/104 | 0/100
Hypothermia (General disorders) | 2/104 | 2/100
Injection Site Erythema (General disorders) | 0/104 | 2/100
Injection Site Phlebitis (General disorders) | 4/104 | 2/100
Injection Site Swelling (General disorders) | 1/104 | 2/100
Oedema (General disorders) | 1/104 | 2/100
Oedema Peripheral (General disorders) | 4/104 | 2/100
Pyrexia (General disorders) | 5/104 | 6/100
Jaundice (Hepatobiliary disorders) | 0/104 | 2/100
Bacteraemia (Infections and infestations) | 3/104 | 2/100
Empyema (Infections and infestations) | 1/104 | 2/100
Pneumonia (Infections and infestations) | 2/104 | 4/100
Staphylococcal Bacteraemia (Infections and infestations) | 3/104 | 4/100
Urinary Tract Infection (Infections and infestations) | 3/104 | 2/100
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0/104 | 2/100
Alanine Aminotransferase Increased (Investigations) | 4/104 | 7/100
Aspartate Aminotransferase Increased (Investigations) | 6/104 | 9/100
Blood Albumin Decreased (Investigations) | 2/104 | 2/100
Blood Alkaline Phosphatase Increased (Investigations) | 12/104 | 9/100
Blood Bilirubin Increased (Investigations) | 3/104 | 2/100
Blood Calcium Decreased (Investigations) | 1/104 | 2/100
Blood Calcium Increased (Investigations) | 0/104 | 2/100
Blood Chloride Increased (Investigations) | 0/104 | 3/100
Blood Creatinine Increased (Investigations) | 3/104 | 3/100
Blood Glucose Decreased (Investigations) | 3/104 | 1/100
Blood Glucose Increased (Investigations) | 1/104 | 3/100
Blood Magnesium Decreased (Investigations) | 4/104 | 4/100
Blood Phosphorus Decreased (Investigations) | 2/104 | 2/100
Blood Potassium Decreased (Investigations) | 6/104 | 8/100
Blood Potassium Increased (Investigations) | 2/104 | 4/100
Blood Sodium Decreased (Investigations) | 1/104 | 3/100
Blood Sodium Increased (Investigations) | 2/104 | 4/100
Blood Urea Increased (Investigations) | 4/104 | 1/100
Blood Uric Acid Decreased (Investigations) | 0/104 | 2/100
Carbon Dioxide Decreased (Investigations) | 0/104 | 2/100
White Blood Cell Count Increased (Investigations) | 1/104 | 3/100
Hyperglycaemia (Investigations) | 2/104 | 3/100
Hypoglycaemia (Investigations) | 1/104 | 3/100
Hypokalaemia (Investigations) | 2/104 | 2/100
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/104 | 3/100
Back Pain (Musculoskeletal and connective tissue disorders) | 1/104 | 2/100
Convulsion (Nervous system disorders) | 3/104 | 0/100
Headache (Nervous system disorders) | 5/104 | 4/100
Agitation (Psychiatric disorders) | 3/104 | 3/100
Confusional State (Psychiatric disorders) | 3/104 | 2/100
Delirium (Psychiatric disorders) | 0/104 | 2/100
Depression (Psychiatric disorders) | 3/104 | 1/100
Insomnia (Psychiatric disorders) | 3/104 | 1/100
Renal Failure (Renal and urinary disorders) | 3/104 | 2/100
Renal Failure Acute (Renal and urinary disorders) | 0/104 | 2/100
Vaginal Discharge (Reproductive system and breast disorders) | 3/104 | 1/100
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1/104 | 2/100
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4/104 | 3/100
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0/104 | 2/100
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2/104 | 2/100
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0/104 | 2/100
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0/104 | 2/100
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 3/104 | 1/100
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 3/104 | 5/100
Pruritus (Skin and subcutaneous tissue disorders) | 0/104 | 3/100
Rash (Skin and subcutaneous tissue disorders) | 5/104 | 3/100
Haematoma (Vascular disorders) | 3/104 | 0/100
Hypertension (Vascular disorders) | 5/104 | 6/100
Hypotension (Vascular disorders) | 7/104 | 3/100
Jugular Vein Thrombosis (Vascular disorders) | 0/104 | 2/100
Phlebitis (Vascular disorders) | 3/104 | 1/100
Venous Thrombosis Limb (Vascular disorders) | 0/104 | 3/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.